CLINICAL TRIAL: NCT06897657
Title: Retrospective, Non-interventional Study of Multiple Sclerosis Routine Clinical Practice: Impact on Adherence and Clinical Outcomes of Ofatumumab Treated Patients
Brief Title: A Study of Multiple Sclerosis Routine Clinical Practice: Impact on Adherence and Clinical Outcomes of Ofatumumab Treated Patients
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: COMB157GGB01
Record Dates: First submitted 2025-03-20; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Disease modifying therapy; Medication adherence; Ofatumumab
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Medication Adherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (3):
- Overall MS Cohort: Adult patients with relapsing-remitting multiple sclerosis (RMS) who were prescribed ofatumumab from either an MS clinic participating in the Kesimpta Connect (KC) patient support program (PSP) or an MS clinic not participating in the KC PSP.
- KC PSP User Cohort: Adult patients with RMS who were prescribed ofatumumab from an MS clinic participating in the KC PSP.
- Non-KC PSP User Cohort: Adult patients with RMS who were prescribed ofatumumab from an MS clinic not participating in the KC PSP.

SUMMARY:
This was a retrospective non-interventional study (NIS) of adult (≥18 years) multiple sclerosis (MS) patients on ofatumumab therapy in the United Kingdom (UK) using secondary data. UK MS centers with National Health Service (NHS) databases and/or homecare and pharmacy services prescribing ofatumumab were identified and recruited for study participation using a feasibility assessment exercise. The study index identification window spanned from 26 March 2021 to 30 June 2023 (or latest data available prior to start of study data extraction). The index date was defined as the first date ofatumumab was dispensed or injected within the index identification window. From index date, patients were followed up until death, up to 13 months after index date, loss to follow-up, or end of study index identification window (whichever came first).

For patients who consented to the use of their data, participating sites transcribed protocol required patient data from existing individual patient medical records into an electronic case report form (eCRF). The end of study was defined as the date of last data query resolution (i.e., all data had been recorded in the eCRF and all data queries resolved to allow database lock to occur). This ensured that all data was available to answer the research questions in the study.

ELIGIBILITY:
Inclusion criteria:

Patients were included in the study if they met all of the following criteria:

* Patient was prescribed ofatumumab within the UK approved marketing authorization
* Patient initiated ofatumumab via participating MS clinic with or without KC PSP
* Patients initiated ofatumumab during the index identification window
* Authorized to collect study data:

  1. Patient was alive at start of data collection and patient consented prior to start of their data collection or,
  2. Patient was deceased at start of data collection and a member of the patient's direct care team had a pre-existing right to access patient medical record
* Specifically for adherence analyses: Patients were required to have a minimum of 6 months of follow-up post index date available to make this assessment
* Specifically for clinical effectiveness analyses: Patients were required to have a minimum of 6 months look-back pre-index date and minimum 6 months follow-up post index date available to make this assessment.

Exclusion criteria:

Patients were excluded from the study if they met the following criteria:

• Patient prescribed ofatumumab outside the approved marketing authorization (i.e., under off-label prescribing) at any point within the patients record

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, non-interventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2023-11-06 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
Medical Possession Ratio (MPR) | Up to 13 months
  MPR was reported as the number of days covered by ofatumumab injections in a given time period, divided by the number of days in the time period.
Number of Patients by MPR Category | Up to 13 months
  MPR was reported as the number of days covered by ofatumumab injections in a given time period, divided by the number of days in the time period. MPR categories:
  * High MPR: MPR = 1.0
  * Intermediate MPR: 0.8 ≤ MPR <1.0
  * Low MPR: MPR <0.8.

SECONDARY OUTCOMES:
Number of Patients by Demographic Category | Baseline
  Demographic categories included:
  * Age group
  * Gender
  * Ethnicity
  * Socioeconomic status (most deprived to least deprived)
  * Decade of MS diagnosis
  * Prior disease modifying treatment (DMT) treatment status (treatment naïve or received prior DMT)
Time From MS Diagnosis to Ofatumumab Initiation | Baseline
Number of Patients by Comorbidity | Baseline
Number of Patients who Received at Least one DMT Prior to Ofatumumab Initiation | Up to 13 months
Number of Prior DMTs Reported | Up to 13 months
Number of Patients by Prior DMT Category | Up to 13 months
  DMT categories included:
  * Type of prior DMT
  * Efficacy of DMT (moderate efficacy, more effective, high efficacy)
  * Use of injectable DMT
  * Type of injectable DMT
Number of Patients by Reason for Switch from Other DMT to Ofatumumab | Up to 13 months
Individual Annualized Relapse Rate (ARR) Before Ofatumumab Initiation | Up to 13 months
  Individual ARR was derived per patient as [(number of confirmed MS relapses) / (time at risk (years)].
Total ARR Before Ofatumumab Initiation | Up to 13 months
  Total ARR was derived as [(total number of confirmed MS relapses) / (total number of person-years at risk)].
Individual ARR After Ofatumumab Initiation | Up to 13 months
  Individual ARR was derived per patient as [(number of confirmed MS relapses) / (time at risk (years)].
Total ARR After Ofatumumab Initiation | Up to 13 months
  Total ARR was derived as [(total number of confirmed MS relapses) / (total number of person-years at risk)].
Average Expanded Disability Status Scale (EDSS) Score Before Ofatumumab Initiation | Up to 13 months
  The EDSS is a tool used to measure how much a person is affected by their MS. It consists of 8 functional systems (FS): Visual, Brain Stem, Pyramidal, Cerebellar, Sensory, Bowel and Bladder, Cerebral and Other functions. Based on the assessment of each FS, the patients score is determined between 0 (normal) and 10 (death due to MS).
Average EDSS Score After Ofatumumab Initiation | Up to 13 months
  The EDSS is a tool used to measure how much a person is affected by their MS. It consists of 8 functional systems (FS): Visual, Brain Stem, Pyramidal, Cerebellar, Sensory, Bowel and Bladder, Cerebral and Other functions. Based on the assessment of each FS, the patients score is determined between 0 (normal) and 10 (death due to MS).
Absolute Change in Average EDSS Score | Up to 26 months
  Absolute change in average EDSS score between 2 study periods was derived as: [mean EDSS score during the follow-up period] - [mean EDSS score during the pre-index period]. The index date was defined as the first date ofatumumab was dispensed or injected within the index identification window.
  The EDSS is a tool used to measure how much a person is affected by their MS. It consists of 8 functional systems (FS): Visual, Brain Stem, Pyramidal, Cerebellar, Sensory, Bowel and Bladder, Cerebral and Other functions. Based on the assessment of each FS, the patients score is determined between 0 (normal) and 10 (death due to MS).
Average Number of T1 and T2 Lesions Before Ofatumumab Initiation | Up to 13 months
Average Number of T1 and T2 Lesions After Ofatumumab Initiation | Up to 13 months
Individual ARR After Ofatumumab Initiation by MPR Category | Up to 13 months
  Individual ARR was derived per patient as [(number of confirmed MS relapses) / (time at risk (years)].
  MPR was reported as the number of days covered by ofatumumab injections in a given time period, divided by the number of days in the time period. MPR categories:
  * High MPR: MPR = 1.0
  * Intermediate MPR: 0.8 ≤ MPR <1.0
  * Low MPR: MPR <0.8.
Total ARR After Ofatumumab Initiation by MPR Category | Up to 13 months
  Total ARR was derived as [(total number of confirmed MS relapses) / (total number of person-years at risk)].
  MPR was reported as the number of days covered by ofatumumab injections in a given time period, divided by the number of days in the time period. MPR categories:
  * High MPR: MPR = 1.0
  * Intermediate MPR: 0.8 ≤ MPR <1.0
  * Low MPR: MPR <0.8.
Average EDSS Score Before Ofatumumab Initiation by MPR Category | Up to 13 months
  The EDSS is a tool used to measure how much a person is affected by their MS. It consists of 8 functional systems (FS): Visual, Brain Stem, Pyramidal, Cerebellar, Sensory, Bowel and Bladder, Cerebral and Other functions. Based on the assessment of each FS, the patients score is determined between 0 (normal) and 10 (death due to MS).
  MPR was reported as the number of days covered by ofatumumab injections in a given time period, divided by the number of days in the time period. MPR categories:
  * High MPR: MPR = 1.0
  * Intermediate MPR: 0.8 ≤ MPR <1.0
  * Low MPR: MPR <0.8.
Average EDSS Score After Ofatumumab Initiation by MPR Category | Up to 13 months
  The EDSS is a tool used to measure how much a person is affected by their MS. It consists of 8 functional systems (FS): Visual, Brain Stem, Pyramidal, Cerebellar, Sensory, Bowel and Bladder, Cerebral and Other functions. Based on the assessment of each FS, the patients score is determined between 0 (normal) and 10 (death due to MS).
  MPR was reported as the number of days covered by ofatumumab injections in a given time period, divided by the number of days in the time period. MPR categories:
  * High MPR: MPR = 1.0
  * Intermediate MPR: 0.8 ≤ MPR <1.0
  * Low MPR: MPR <0.8.
Absolute Change in Average EDSS Score by MPR Category | Up to 26 months
  Absolute change in average EDSS score between 2 study periods was derived as: [mean EDSS score during the follow-up period] - [mean EDSS score during the pre-index period]. The index date was defined as the first date ofatumumab was dispensed or injected within the index identification window.
  The EDSS is a tool used to measure how much a person is affected by their MS. It consists of 8 functional systems (FS): Visual, Brain Stem, Pyramidal, Cerebellar, Sensory, Bowel and Bladder, Cerebral and Other functions. Based on the assessment of each FS, the patients score was determined between 0 (normal) and 10 (death due to MS).
  MPR was reported as the number of days covered by ofatumumab injections in a given time period, divided by the number of days in the time period. MPR categories:
  * High MPR: MPR = 1.0
  * Intermediate MPR: 0.8 ≤ MPR <1.0
  * Low MPR: MPR <0.8.
Number of Patients per MPR Category by Type of KC PSP Services Received | Up to 13 months
  KC PSP services included face-to-face nurse visits, virtual nurse visits, and mobile text reminders.
  MPR was reported as the number of days covered by ofatumumab injections in a given time period, divided by the number of days in the time period. MPR categories:
  * High MPR: MPR = 1.0
  * Intermediate MPR: 0.8 ≤ MPR <1.0
  * Low MPR: MPR <0.8.
Number of Medical Visits After Ofatumumab Initiation | Up to 13 months
  Medical visits included accident and emergency (A&E) visits, inpatient visits, and outpatient visits.
Annualized Medical Visit Rate After Ofatumumab Initiation | Up to 13 months
  Annualized medical visit rate per patient was calculated as [(number of events during follow-up period) / (time at risk (years) during follow-up period)]. Rates were calculated for the following types of medical visits: A&E visits, inpatient visits, and outpatient visits.
Number of MS-related Medical Visits After Ofatumumab Initiation | Up to 13 months
  MS-related medical visits included A&E visits, inpatient visits, and outpatient visits.
Annualized MS-related Medical Visit Rate After Ofatumumab Initiation | Up to 13 months
  Annualized MS-related medical visit rate per patient was calculated as [(number of events during follow-up period) / (time at risk (years) during follow-up period)]. Rates were calculated for the following types of MS-related medical visits: A&E visits, inpatient visits, and outpatient visits.
Number of Patients With Medically Reported Adherence (MRA) After Ofatumumab Initiation | Up to 13 months
  Full adherence was defined as no record of dose/s missed between ofatumumab initiation and the point at which the patient was censored. Partial adherence was defined as a record of at least one dose missed between ofatumumab initiation and the point at which the patient was censored. The date of censoring was defined as the earliest of the following:
  * End of the study follow-up (13 months)
  * Death
  * Lost to follow-up
  * End of study index identification period
Number of Patients by Reason for Discontinuation of Ofatumumab | Up to 13 months
Number of Patients who Switched From Ofatumumab to an Alternative DMT | Up to 13 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States